CLINICAL TRIAL: NCT02743065
Title: Superselective Drug-Eluting Chemoembolization With HepaSphere in Unresectable Advanced HCC Patients: Safety & Efficacy Registry in China (SUPER-China)
Brief Title: HepaSphere Chemoembolization in Advanced HCC Patients: Safety & Efficacy Registry in China
Acronym: SUPER-China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hong Shan, Professor, Fifth Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: HEPA-China-002
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: HepaSphere
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Device: HepaSphere Microspheres: HepaSphere Microsphere
  Interventions: Device: HepaSphere with 50-75mg Doxorubicin

INTERVENTIONS:
Device: HepaSphere with 50-75mg Doxorubicin — HepaSphere with 50-75mg Doxorubicin
  Other Names: Superaborbent Polymer Microsphere

SUMMARY:
The purpose of this multicenter registry is to gather the safety, efficacy and survival data in advanced HCC patients treated with HepaSphere in China in order to evaluate the application of HepaSphere deTACE in treating advanced HCC patients

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Patient has signed informed consent
3. Patient must have a diagnosis of hepatocellular cancer by at least one of the following method:

   1. Histological confirmation
   2. Classic imaging characteristics of HCC: Early enhancement (Arterial hypervascularity) and Venous or Delayed phase washout in multidetector contrast enhanced computed tomography (CT) scan / dynamic contrast-enhanced magnetic resonance imaging (MRI) imaging.

      * Either CT/ MRI shows at least one solid liver lesion ≥ 2 cm with the above described imaging characteristics of HCC.
      * In case of liver lesion between 1 and 2 cm, both CT and MRI imaging have to be performed in order to confirm the imaging characteristics of HCC.
4. At time of study entry.

   1. Patients not suitable for ablation due to lesion location may be enrolled
   2. Patients with HCC recurrence but not suitable for resection or ablation maybe enrolled
5. Patient MUST be with BCLC stage C and meet the following criteria:

   * Stage Child-Pugh A or B AND
   * Performance status ECOG ≤ 2 WITH Vascular Invasion or WITHOUT Vascular invasion
6. Patient has a life expectancy of at least 6 months

Exclusion Criteria:

1. Current or previous treatment with chemo- or radiation therapy or sorafenib
2. Previous treatment of transarterial chemoembolization (TACE)
3. Patients with current or history of any other cancer except non-melanomatous skin cancer
4. Female patients who are pregnant, breastfeeding, or premenopausal and not using an effective method of contraceptive
5. Performance status ECOG > 2
6. Child-Pugh Class C
7. Occlusive tumor thrombus to the main portal trunk
8. Active gastrointestinal bleeding
9. Evidence of uncorrectable bleeding diathesis
10. Extra-Hepatic spread of the HCC
11. >50% tumor involvement of the liver
12. Infiltrative HCC
13. Encephalopathy not adequately controlled medically
14. Presence of ascites not controlled medically
15. Any contraindication for MRI/ CT (eg. metallic implants)
16. Allergy to contrast media that cannot be managed with prophylaxis
17. Any contraindication to arteriography
18. Any contraindication for doxorubicin administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Advanced Hepatocellular Carcinoma (HCC)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 2- years
Progress-free-survival (PFS) | 2-years

SECONDARY OUTCOMES:
Overall Survival | 2-years
Objective Response Rates | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Hong Shan, MD, Principal Investigator — Fifth Affiliated Hospiatl, Sun Yet-Sen University
Locations (6):
- China (6):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Fifth Affiliated Hospiatl, Sun Yet-Sen University, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Third Affiliated Hospiatl, Sun Yet-Sen Hospital, Guangzhou
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided